CLINICAL TRIAL: NCT00616460
Title: ACRIPAB- Trial: Anti Coagulation Regimen In High Risk PAtients for Bleeding
Acronym: ACRIPAB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Turgeman Yoav, Chief of Cardiology Department, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0124-07-EMC
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Hematologic Diseases
Keywords: safety; efficacy
MeSH Terms: conditions — Hematologic Diseases | interventions — bivalirudin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bivalirudin (Experimental)
  Interventions: Drug: Bivalirudin

INTERVENTIONS:
Drug: Bivalirudin — Bivalirudin: loading dose 0.75mg/kg bolus During procedure: 1.75mg/kg/hour. UFH: loading dose 60 Units /kg During procedure: keeping ACT < 250

SUMMARY:
To determine the safety/efficacy of Bivallirudin Vs unfractionated heparin (UFH) on top of dual antiplatelet therapy in patients with high tendency for bleeding during urgent and elective PCI.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria (any of the following):

* ≥75 years
* Creatinin clearance rate < 60 ml per minute
* Anemia (Hb 9-11 mg%)
* Hypertension: BP > 180/95 mmHg but less than 210/110 m Hg
* Diabetic Pts
* Steroid treated Pts
* Recent (within 6 weeks) non major surgery
* Pts with hematological disorders associated with tendency for bleeding like Thrombocytopenia (platelets 50000-150000) included TTP;

Exclusion Criteria:

Exclusion criteria:

* Age < 18 year
* Acute STEMI (Primary PCI)*
* Rescue angioplasty <12h after lytic therapy*
* Active bleeding
* S.C LMWH < 8 hours or UFH < 4 hours before PCI
* Using IIb /IIIa as an upstream therapy before PCI
* PCI which will be involved with obligatory IIb /IIIa therapy:

(thrombotic complication, occlusive dissection)

* INR>1.5 on day of cathetrization
* Bolus of 600mg of Clopidogrel before PCI
* Current pregnancy or women in reproductive age without contraceptives
* Hypersensitivity to heparin or bivalirudin or its components *(possible using IIB/IIIA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
End points: Primary :Major & minor bleeding Port of entry related complications | 30 days

SECONDARY OUTCOMES:
End points: Secondary: 30 days MACE | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Turgeman, MD, Principal Investigator — Heart Institute HaEmek medical center
Locations (1):
- Heart Institute haEmek Medical Center, Afula, Israel